CLINICAL TRIAL: NCT02121626
Title: The FOCCUS Study: "Focusing on Cancer Chemotherapys' Untreated Symptoms"
Brief Title: The FOCCUS Study: "Focusing on Cancers Chemotherapys' Untreated Symptoms"
Acronym: FOCCUS
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR 3921
Record Dates: First submitted 2014-04-17; First posted 2014-04-23 (Estimated); Last update posted 2017-11-22 (Actual); Status verified 2017-11

CONDITIONS: Cancer
Keywords: Cancer; Chemotheraphy; Small Bowel Bacterial Overgrowth; Bile Acid Malabsorption; Pancreatic Insufficiency; Carbohydrate Malabsorption; Anorexia; Borborygmi; Bloating; Constipation; Diarrhoea; Mucositis; Dysphagia; Early satiety; Frequency of defaecation; Incontinence; Mucus discharge; Nausea; Nocturnal defaecation; Pain; Reflux; Regurgitation; Steatorrhoea; Tenesmus; Urgency of defaecation; Vomiting; Weight loss; Wind.
MeSH Terms: conditions — Neoplasms; Exocrine Pancreatic Insufficiency; Anorexia; Constipation; Diarrhea; Mucositis; Deglutition Disorders; Nausea; Pain; Gastroesophageal Reflux; Steatorrhea; Vomiting; Weight Loss; Flatulence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and Stool Samples will be collected for translational analysis.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Chemotheraphy Treatement: The study will be limited to NHS patients to reduce complications associated with the need for additional funding authorisations from private health care providers for algorithm-instigated investigations. It is not envisaged that participation in other studies running within the GI unit at The Royal Marsden Hospital will preclude entry into this study except in the event of those rare studies where the study is specifically measuring toxicity of treatment as the primary end point.

SUMMARY:
The aim of the study is to identify how often gastrointestinal problems interfere with quality of life as a result of treatment for cancer with chemotherapy. We also want to identify the causes for these symptoms and see if simple treatments used for other gastrointestinal conditions could make chemotherapy an easier experience. Chemotherapy for cancer can be hard work for the patient. Often it makes them feel tired. Not infrequently, it can cause a whole range of physical side effects. Probably the most common side effects are those affecting the stomach and bowels. Vomiting used to be a major problem with chemotherapy but research discovered a whole series of new treatments so that severe vomiting from chemotherapy is rarely a problem today. However, patients can develop a whole series of other symptoms during chemotherapy, for example, bloating, wind, diarrhoea, needing to rush to the lavatory and opening the bowels very frequently. The causes for these symptoms have hardly been studied even though they sometimes affect people quite badly. In our specialist gastrointestinal clinic at the Royal Marsden Hospital, over the last 12 years, we have pioneered new methods for dealing with symptoms which affect the bowel after radiotherapy. We would like to extend these methods to people having chemotherapy. We have identified several easily treatable causes for these symptoms after radiotherapy, which previously were often ignored. We believe that some of these causes also occur in people having chemotherapy and if we knew how often they do occur we could focus on improving treatment for affected people. We plan to find out how often 40 stomach and bowel symptoms occur during chemotherapy. In people who are troubled by any or some of these symptoms we will arrange simple series tests which could sort out why these symptoms occur and we will record how they respond to treatment.

DETAILED DESCRIPTION:
Chemotherapy (CT) remains an integral part of treatment for many types of cancer often in combination with surgery and/or radiotherapy. In the year March 2011 to April 2012, 1807 patients were referred to the Royal Marsden Hospital (RMH) Gastrointestinal Unit with a new gastro intestinal (GI) cancer of whom 709 were treated with chemotherapy alone or in combination with other long term outcome. GI symptoms are common in patients receiving chemotherapy. They may arise from the tumour, but may also result as a side effect of treatment. They include anorexia, borborygmi, bloating, constipation, diarrhoea, dysphagia, early satiety, frequency of defaecation, incontinence, mucus discharge, nausea, nocturnal defaecation, pain, reflux, regurgitation, steatorrhoea, tenesmus, urgency of defaecation, vomiting, weight loss and wind. Frequently, such symptoms have a significant impact on patients' quality of life. They may also interfere with the delivery of treatment prompting cessation of therapy or dose reduction resulting in sub optimal dosage with a potential impact on morbidity and mortality. Whilst clinicians have long focused on the management of vomiting and pain in cancer patients, less attention has been paid to the incidence, severity or optimal management of other GI symptoms. If the cause of these symptoms can be identified, then appropriate investigations and treatments can be prescribed. The GI Unit has successfully investigated and treated patients with symptoms emerging after radiotherapy. This experience has enabled the team to develop an algorithm for facilitating the investigation and treatment of cancer therapy induced symptoms. The algorithm has recently been shown to be effective in the management of patients with radiation induced bowel injury . In particular, it enables the rapid identification of required investigations and improves the management of symptoms that might otherwise be mislabeled as inevitable consequences of treatment. Five easily treatable causes for GI symptoms have so far been identified:

* Small bowel bacterial overgrowth
* Carbohydrate malabsorption
* Bile acid malabsorption
* Gastric bile reflux
* Pancreatic insufficiency

It is likely that additional causes such as viral infections (eg cytomegalovirus) are more frequent in patients undergoing chemotherapy than currently appreciated.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above able to give informed consent
* Patients referred to one of the five prescribing consultants described above
* Patients to be treated within the GI unit at the Royal Marsden Hospital (RMH Chelsea, Sutton or Kingston) with chemotherapy with or without other treatments.

Exclusion Criteria:

* Patients aged less than 18 years
* Patients unable to give informed consent
* Patients being treated privately
* Patients on studies with conflicting end-points

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at The Royal Marsden NHS Foundation Trust who have been diagnosed with cancer and are receiving chemotherapy as part of their treatment. This study will recruit men and women who will receive chemotherapy for cancers of the oesophagus, stomach, pancreas, liver, biliary tree or bowel.
Sampling Method: Non-Probability Sample
Enrollment: 248 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Incidence of new onset GI symptoms per chemotherapy regimen | Every 4 weeks

SECONDARY OUTCOMES:
Change in Gastrointestinal Symptom Rating Scale (GSRS) scores | Every 4 weeks
Change in Vaizey incontinence scores | Every 4 weeks
Change in Bristol Stool Chart parameters (stool frequency, type, mode) | Every 4 weeks
Change in Quality of Life scores (FACTG, version 4 questionnaires) | Every 4 weeks
Change in neurotoxicity scores (FACT/GOGNTX13, version 4) | Every 4 weeks
Competency (learning outcomes) GI research nurses | Every 2 months
Identification of genetic profiles which predispose to specific chemotherapy induced toxicities. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jervoise Andreyev, MBBS, Ph.D, Study Chair — Royal Marsden NHS Foundation Trust; Linda Wedlake, RD MSc BSc, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- The Royal Marsden NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Andreyev HJN, Lalji A, Mohammed K, Muls ACG, Watkins D, Rao S, Starling N, Chau I, Cruse S, Pitkaaho V, Matthews J, Caley L, Pittordou V, Adams C, Wedlake L. The FOCCUS study: a prospective evaluation of the frequency, severity and treatable causes of gastrointestinal symptoms during and after chemotherapy. Support Care Cancer. 2021 Mar;29(3):1443-1453. doi: 10.1007/s00520-020-05610-x. Epub 2020 Jul 16. PMID 32676853